CLINICAL TRIAL: NCT03840473
Title: Efficacy of Combination Therapies on Neck Pain and Muscle Tenderness in Patients With Upper Trapezius Myofascial Trigger Points
Brief Title: Efficacy of Combination Therapies on Neck Pain & Muscle Tenderness in Patients With Upper Trapezius MTrPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Collaborators: Shah Physiotherapy Center, Delhi, India (Unknown)
Responsible Party: Principal Investigator, AMIR IQBAL, Principle Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRC-2017-007
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Myofascial Trigger Point Pain
Keywords: Neck pain; Upper trapezius muscle; Myofascial trigger points; Muscle tenderness; Pain pressure threshold
MeSH Terms: conditions — Myofascial Pain Syndromes; Neck Pain; Myalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MET+ICT+Conventional intervention (Experimental): Hot packs (75°C) for 20 minutes and supervised active stretching exercises for upper trapezius muscle (slow, 5 repetitions per session, 10-second hold and 10-second relaxation between two repetitions) followed by ICT (90-second hold-time) and MET (5-second hold-time, 3-second relaxation by exhalation while reaching the new barrier).
  Interventions: Behavioral: MET; Behavioral: ICT; Behavioral: Conventional Intervention
- MET+Conventional Intervention (Experimental): Hot packs (75°C) for 20 minutes and supervised active stretching exercises for upper trapezius muscle (slow, 5 repetitions per session, 10-second hold and 10-second relaxation between two repetitions) followed by MET (5-second hold-time, 3-second relaxation by exhalation while reaching the new barrier).
  Interventions: Behavioral: MET; Behavioral: Conventional Intervention
- Conventional Intervention (Active Comparator): Received hot packs (75°C) for 20 minutes and supervised active stretching exercises for upper trapezius muscle (slow, 5 repetitions per session, 10-second hold and 10-second relaxation between two repetitions) only.
  Interventions: Behavioral: Conventional Intervention

INTERVENTIONS:
Behavioral: MET — The patient was in a supine position with the cervical spine in the opposite lateral flexion to the treating part so that the upper trapezius muscle fibers were in a lengthened position.19 The moderate isometric contraction (approximately 75% of maximal) of the upper trapezius muscles was elicited for a period of 5 seconds followed by 3 seconds of relaxation while reaching the new barrier. The technique was repeated four times in each session.
  Arms: MET+Conventional Intervention; MET+ICT+Conventional intervention
Behavioral: ICT — The patient lying in the supine position with the cervical spine in opposite lateral flexion to the treating part so that the upper trapezius muscle fibers were kept in a lengthened position.18,22 The physiotherapist applied gradually increasing pressure to the MTrPs until the subject perceived the first noticeable pain. At that moment, the pressure was maintained until the discomfort and/or pain eased by around 50% as perceived by the patient, at which time the pressure was increased until the discomfort appeared again. This process was maintained for 90 seconds.
  Arms: MET+ICT+Conventional intervention
Behavioral: Conventional Intervention — Hot packs (75°C) for 20 minutes and active stretching exercises for the upper trapezius muscle (slow, 5 repetitions per session, 10-second hold and 10-second relaxation between two repetitions). Active stretching exercises were done by all the participants under the supervision of the physical therapist. This approach was standardized for all participants.

SUMMARY:
Myofascial pain syndrome thought to be the main cause of neck pain and shoulder muscle tenderness in the working population is characterized by myofascial trigger points (MTrPs). This study aimed to examine the immediate and short-term effect of the combination of two therapeutic techniques for improving neck pain and muscle tenderness in patients with upper trapezius Myofascial Trigger points.

DETAILED DESCRIPTION:
Purpose: Myofascial pain syndrome, thought to be the main cause of neck pain and shoulder muscle tenderness in the working population, is characterized by myofascial trigger points (MTrPs). This study aimed to examine the immediate and short-term effect of the combination of two therapeutic techniques for improving neck pain and muscle tenderness in male patients with upper trapezius active MTrPs.

Methods: This was a pretest-posttest single-blinded randomized controlled trial. Sixty male subjects with mechanical neck pain due to upper trapezius active MTrPs were recruited and randomly allocated into group A, which received muscle energy technique (MET) and ischemic compression technique (ICT)along with conventional intervention; group B, which received all the interventions of group A except ICT; and group C, which received conventional treatment only. Baseline (Pr), immediate post-intervention (Po), and 2-week follow-up (Fo) measurements were made for all variables. Pain intensity and pressure pain threshold (PPT)were assessed by a visual analog scale (VAS) and pressure threshold meter, respectively. All three groups received their defined intervention plans only. Repeated-measures analysis of variance was used to perform intra- inter-group analyses. Cohen's d test was used to assess the effect size of the applied interventions within the groups.

ELIGIBILITY:
Inclusion Criteria:

* Male subject diagnosed with non-specific neck pain and muscle tenderness over the upper trapezius muscle due to an active MTrP
* Age19-38 years
* Presence of a maximum of 1-2active MTrPs in a unilateral upper trapezius muscle The number of TrPs in upper trapezius is not limited to two; it may be one or may be more than two (satellite TrPs) also. However, due to time constraints of the study sessions allowed for treatment of up to 2 active MTrPs only.

Exclusion Criteria:

* Diagnosed with fibromyalgia syndrome according to the American College of Rheumatology criteria;
* Had active MTrPs in the bilateral upper trapezius muscles
* Had a history of whiplash injury or cervical spine surgery
* Were diagnosed with cervical radiculopathy or myelopathy determined by their primary health care physician
* Had accepted myofascial pain therapy within the 1 month before the study
* Showed poor cooperation.

Ages: 19 Years to 38 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male only
Enrollment: 60 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2017-12-19 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Muscle tenderness | Change from baseline PPT scores at day 1 post intervention and after 2-weeks follow-up
  A pressure algometer used to assess the muscle tenderness by measuring Pressure Pain Threshold (PPT) level of MTrPs as suggested by Fischer. The trigger point with the lowest PPT value was chosen as a primary trigger point. The subjects were instructed to indicate the sensation of pressure they felt from changing from one of pressure to one of pain by saying "there"/ "yes." Three repeated measurements were obtained by the same assistant, and the mean was used in the analysis. At least a 1-minute gap was added between the two repeated measurements as recommended by Fischer.
Neck pain intensity | Change from baseline VAS scores at day 1 post intervention and after 2-weeks follow-up
  Visual analogue scale (VAS) used to measure neck pain intensity. VAS is a subjective rating scale marked with 0 (No pain) and 10 (extremely unbearable pain) on its either end. An application of 2.5 kg/cm-square of pressure was applied at the rate of 1 kg/cm-square by the physiotherapist while the subjects were stated to rate their pain on the visual analog scale (VAS) to evaluate local pain evoked by the application of that amount of pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Iqbal, MPT, Principal Investigator — Rehabilitation Research Chair
Locations (1):
- Rehabilitation Research Chair, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided